CLINICAL TRIAL: NCT06403982
Title: The Influence of Oxytocin on Intrapartum Fetal Well-being and Delivery Outcomes in Patients Receiving Epidural Analgesia - a Randomized Controlled Trial
Brief Title: The Influence of Oxytocin on Intrapartum Fetal Well-being and Delivery Outcomes in Patients Receiving Epidural Analgesia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Król Joanna, Principal Investigator, MD, Central Clinical Hospital of the Ministry of Internal Affairs and Administration, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KB 26/2024
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Uterine Contraction; Oxytocin; Labor Progress; Fetal Doppler; Labor Epidural Analgesia; Labor Pain
Keywords: epidural anaesthesia; use of oxytocin; uterine contractions; fetal well-being; fetal doppler; ctg; fetal monitoring; labor analgesia; labor pain; labor progression
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin Group (Experimental): Oxytocin Group will comprise 100 women in labor either stimulated or induced by oxytocin requesting epidural analgesia (ELA). The use of oxytocin will be continued after the administration of ELA.
  Interventions: Other: Continuation of oxytocin after ELA
- Control Group (Placebo Comparator): Control Group will comprise 100 women in labor either stimulated or induced by oxytocin requesting epidural analgesia (ELA). The oxytocin pump will be changed to 0.9% sodium chloride solution pump after the administration of ELA.
  Interventions: Other: Discontinuation of oxytocin after ELA

INTERVENTIONS:
Other: Continuation of oxytocin after ELA — The use of oxytocin will be continued after the administration of ELA. The vital signs (blood pressure, saturation, heart rate) and the Doppler velocities in the uterine arteries, umbilical artery and the fetal middle cerebral artery will be measured directly before the administration of ELA and then after 30, 60 and 120 minutes. After 2 hours the patients will be examined to assess the progress of labor.
  Additionally, the velocities in the uterine arteries will be measured during the first day after the delivery.
  Arms: Oxytocin Group
Other: Discontinuation of oxytocin after ELA — The oxytocin pump will be changed to 0.9% sodium chloride solution pump after the administration of ELA. The vital signs (blood pressure, saturation, heart rate) and the Doppler velocities in the uterine arteries, umbilical artery and the fetal middle cerebral artery will be measured directly before the administration of ELA and then after 30, 60 and 120 minutes. After 2 hours the patients will be examined to assess the progress of labor. If no progress is detected due to the secondary weakening of uterus contractile function, the oxytocin will be reintroduced. Additionally, the velocities in the uterine arteries will be measured during the first day after the delivery.
  Arms: Control Group

SUMMARY:
The aim of this study is to determine the influence of oxytocin on fetal well-being during labor in patients receiving epidural analgesia (ELA) with the use of cardiotocography (CTG) and doppler ultrasonography.

CTG is a commonly used technique to monitor the fetal heartbeat and contractions of uterus during pregnancy and labor. The maternal-fetal doppler ultrasonography is a non-invasive method used for the pregnancy surveillance.

Various psychological and psychosocial factors impact the perception of labor pain. Its intensity is described differently by each patient - some claim it to be the worst pain that they experienced during their lives. Usually, the labor pain is more severely experienced by the patients giving birth for the first time and those with induced labor.

Nowadays, there are many non-pharmacological (e.g. acupuncture, massage, TENS) and pharmacological (anesthetic gas, opioids, ELA) methods of labor pain management. ELA is a regional anesthesia, in which the anesthetic drug is injected into the epidural space with the aim to block the pain experienced by the patient without impacting patients ability to move or push during labor. The safety of the procedure is well-discussed and documented in Cochrane review from 2018, which shows no adverse impact on the proportions of Caesarean section, long-term backache, or neonatal outcomes. It is considered to be a golden standard for labor pain management.

Oxytocin is a well-known hormone used for the induction of labor and to stimulate the uterine contraction during labor. The impact of oxytocin alone on CTG pattern and maternal-fetal doppler ultrasonography is discussed in the literature. However, the cumulative effect of ELA and oxytocin remains unclear. Some researchers claim that ELA increases the frequency of uterine contractions and that the additional use of oxytocin leads to higher risk of uterine hyper-stimulation and unreassuring CTG patterns. Whereas the others state that ELA weakens the strength of uterine contractions leading to slow progression of labor and the need to use or increase the use of oxytocin.

There are no data on how the cumulative use of oxytocin and ELA impacts the maternal-fetal flows during labor.

DETAILED DESCRIPTION:
This is a randomized controlled trial performed at the Clinical Department of Obstetrics and Perinatology at the National Medical Institute of the Ministry of the Interior and Administration. The study will recruit 200 patients in either labor induced by oxytocin or stimulated with oxytocin at 37-42 weeks of gestation, requesting the epidural labor analgesia (ELA) and meeting the inclusion criteria. The patients will be individually randomized to either the study group (n=100), in which the use of oxytocin will be continued after the administration of ELA; or to the control group (n=100), in which the oxytocin will be changed to 0.9% sodium chloride solution after the ELA administration.

The vital signs (blood pressure, saturation, heart rate) and the Doppler velocities in the uterine arteries, umbilical artery and the fetal middle cerebral artery will be measured directly before the administration of ELA and then after 30, 60 and 120 minutes. After 2 hours the patients will be examined to assess the progress of labor. If no progress is detected due to the secondary weakening of uterus contractile function, the oxytocin will be reintroduced in the control group.

Additionally, the velocities in the uterine arteries will be measured during the first day after the delivery.

The labor and neonatal outcomes (e.g mode of the delivery, duration of labor, Apgar score, umbilical artery blood gas analysis) will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* singleton pregnancy
* labor induced by oxytocin or stimulated with oxytocin
* signed informed consent form
* cervical dilation ≥ 3cm
* patient requesting and eligible for epidural analgesia
* normal CTG trace for at least 30 minutes before epidural analgesia

Exclusion Criteria:

* less than 18 years old
* preterm delivery
* multiple pregnancy
* fetal malformations
* less than 3cm cervical dilation
* lack of CTG trace for at least 30 minutes before epidural analgesia
* patient not requesting or not eligible for epidural analgesia
* informed consent form not signed
* spontaneous labor without the use of oxytocin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-06 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in CTG pattern | During the first two hours after the enrollment
  E.g. changes in fetal heart rate, presence of cycling, presence of decelerations, STV value in both arms
Maternal-Fetal Doppler | From the enrollment to the first day after the delivery
  The PI values in uterine arteries, umbilical artery and fetal middle cerebral artery
Labour progression | The first two hours after the enrollment
  The change in cervical dilation

SECONDARY OUTCOMES:
Duration of labor | From the enrollment to two hours after the delivery
  Duration of first and second stages of labor
Mode of the delivery | At the time of delivery
  Vaginal Birth or Assisted vaginal birth or Caesarean section
Umbilical cord blood gasometry | At the delivery
  The result of umbilical cord blood gasometry at the delivery
Apgar score | At the delivery of newborn
  Newborn Apgar score in 1, 3 and 5th minute
Birth weight of the newborn | At the delivery
  Birth weight of the newborn
Presence of Neonatal Complications | From the delivery to the hospital discharge of the newborn
  hospitalization at neonatal intensive care unit, infections, respiratory or neurological disorders etc.
Presence of labor complications | From enrollment up to two hours after the delivery
  Lack of labor progress, Postpartum hemorrhage, Fetal distress, Placental abruption etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Department of Obstetrics and Perinatology, National Medical Institute of the Ministry of the Interior and Administration, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on reasonable request
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Study protocol will be available following its publication. The anonymized participant data will become available upon publishing the protocol and the results of the study.
Access Criteria: The data will be provided on reasonable request. (contact details: joanna.krol@wum.edu.pl).
URL: https://szkoladoktorska.wum.edu.pl

REFERENCES:
- [Background] Ye Y, Song X, Liu L, Shi SQ, Garfield RE, Zhang G, Liu H. Effects of Patient-Controlled Epidural Analgesia on Uterine Electromyography During Spontaneous Onset of Labor in Term Nulliparous Women. Reprod Sci. 2015 Nov;22(11):1350-7. doi: 10.1177/1933719115578926. Epub 2015 Mar 29. PMID 25824008
- [Background] Anim-Somuah M, Smyth RM, Cyna AM, Cuthbert A. Epidural versus non-epidural or no analgesia for pain management in labour. Cochrane Database Syst Rev. 2018 May 21;5(5):CD000331. doi: 10.1002/14651858.CD000331.pub4. PMID 29781504
- [Background] Lurie S, Feinstein M, Heifetz C, Mamet Y. Epidural analgesia for labor pain is not associated with a decreased frequency of uterine activity. Int J Gynaecol Obstet. 1999 May;65(2):125-7. doi: 10.1016/s0020-7292(99)00005-3. PMID 10405055
- [Background] Abrao KC, Francisco RPV, Miyadahira S, Cicarelli DD, Zugaib M. Elevation of uterine basal tone and fetal heart rate abnormalities after labor analgesia: a randomized controlled trial. Obstet Gynecol. 2009 Jan;113(1):41-47. doi: 10.1097/AOG.0b013e31818f5eb6. PMID 19104358